CLINICAL TRIAL: NCT01029340
Title: A Two Part Randomized Cross-Over Trial to Evaluate the Pharmacokinetics, Efficacy, and Safety Profile of Plasma Protein-Free Recombinant FVIII Formulated With Sucrose (BAY81-8973) in Previously Treated Subjects With Severe Hemophilia A Under Prophylaxis Therapy
Brief Title: Trial to Evaluate the Efficacy and Safety of a New Full Length Recombinant Human FVIII for Hemophilia A
Acronym: Leopold I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12954; 2009-012149-43 (EudraCT Number)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Blood Coagulation Disorders; Hemophilia A
Keywords: Hemophilia A; Factor VIII; Prophylaxis
MeSH Terms: conditions — Blood Coagulation Disorders; Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1: Recombinant Factor VIII (BAY81-8973) then Kogenate FS (Experimental): Part A - Arm 1: Participants first received one single intravenous (IV) injection of BAY81-8973 50 IU/kg, then 1 single IV injection of Kogenate FS (BAY14-2222) 50 IU/kg with a wash-out period of at least 2-3 days in between
  Interventions: Biological: Recombinant Factor VIII (BAY81-8973)
- Arm 2: Kogenate FS then Recombinant Factor VIII (BAY81-8973) (Experimental): Part A - Arm 2: Participants first received one single intravenous (IV) injection of Kogenate FS (BAY14-2222) 50 IU/kg, then 1 single IV injection of BAY81-8973 50 IU/kg with a wash-out period of at least 2-3 days in between
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)
- Arm 3: Recombinant Factor VIII by CS/EP then by CS/ADJ (Experimental): Part B - Arm 3: Participants received IV injection of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay Potency Per European Pharmacopeia for 6 months and then crossed over to study drug measured by Chromogenic Substrate Assay/Adjusted to Label Potency for 6 months
  Interventions: Biological: Recombinant Factor VIII (BAY81-8973)
- Arm 4: Recombinant Factor VIII by CS/ADJ then by CS/EP (Experimental): Part B - Arm 4:. Participants received IV injection of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay/Adjusted to Label Potency for 6 months and then crossed over to study drug measured by Chromogenic Substrate Assay Per European Pharmacopeia for 6 months
  Interventions: Biological: Recombinant Factor VIII (BAY81-8973)
- Arm 5: Recombinant Factor VIII by CS/EP (Experimental): Part C - Arm 5: Participants received a loading dose of approximately 50 IU/kg of BAY 81-8973 before the first surgical incision followed by further treatment with BAY 81-8973 according to surgical requirements for up to 3 weeks
  Interventions: Biological: Recombinant Factor VIII (BAY81-8973)

INTERVENTIONS:
Biological: Recombinant Factor VIII (BAY81-8973) — Single dose of BAY81-8973 crossed over to single dose of Kogenate FS
  Arms: Arm 1: Recombinant Factor VIII (BAY81-8973) then Kogenate FS
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Single dose of Kogenate FS crossed over to Single dose of BAY81-8973
  Arms: Arm 2: Kogenate FS then Recombinant Factor VIII (BAY81-8973)
Biological: Recombinant Factor VIII (BAY81-8973) — Participants received IV injections of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay Potency Per European Pharmacopeia (CS/EP) for 6 months and by Chromogenic Substrate Assay/Adjusted to Label Potency (CS/ADJ) for 6 months, sequence according to randomization.
  Arms: Arm 3: Recombinant Factor VIII by CS/EP then by CS/ADJ; Arm 4: Recombinant Factor VIII by CS/ADJ then by CS/EP
Biological: Recombinant Factor VIII (BAY81-8973) — Participants received a loading dose of approximately 50 IU/kg of BAY 81-8973 before the first surgical incision followed by further treatment with BAY 81-8973 according to surgical requirements for up to 3 weeks
  Arms: Arm 5: Recombinant Factor VIII by CS/EP

SUMMARY:
The study will assess the pharmacokinetics (part A) safety, tolerability, and efficacy of prophylaxis treatment (2 to 3 times a week) (part B) with BAY81-8973 over a one year period (split into two six month treatment periods). The study will compare 2 different methods (assays) for measuring the amount of study drug, the chromogenic substrate assay per European Pharmacopeia (CS/EP) with the classical assay (Chromogenic Substrate Adjusted, CS/ADJ). During one six month period patients will receive the study drug where the dose has been measured using the" (CS/EP) and during the other six months period the dose will be measured based on the Chromogenic Substrate Adjusted assay CS/ADJ)

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 12 to 65 years
* Severe hemophilia A defined as < 1% FVIII:C
* >/= 150 days of previous treatment with FVIII in lifetime
* Currently receiving on-demand or any type of prophylaxis treatment regimen with any FVIII product
* No history of or current FVIII inhibitors

Exclusion Criteria:

* Presence of another bleeding disease that is different from hemophilia A (e.g., von Willebrand disease, hemophilia B)
* Low platelet count, abnormal kidney function, or liver disease
* Received treatment with immune suppressing drugs within the last 3 months prior or requires treatment during the study. (Some drugs for hepatitis C, Human immunodeficiency virus (HIV), and steroids are allowed)
* Receiving or has received other experimental drugs within 3 months prior to study entry
* Allergy to Factor VIII or hamsters or mouse protein

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (58):
- United States (7):
  - Orange, California
  - Sacramento, California
  - Tampa, Florida
  - Boston, Massachusetts
  - East Lansing, Michigan
  - Kansas City, Missouri
  - Cleveland, Ohio
- Argentina (2):
  - Bahía Blanca, Buenos Aires
  - Rosario, Santa Fe Province
- Austria (2):
  - Vienna, Vienna
  - Graz
- Zagreb, Croatia
- DK-Aarhus N, Denmark
- Germany (5):
  - Frankfurt am Main, Hesse
  - Bonn, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Magdeburg, Saxony-Anhalt
- Hong Kong, Hong Kong
- India (3):
  - Bangalore
  - Mumbai
  - Pune
- Jakarta, Indonesia
- Ramat Gan, Israel
- Italy (5):
  - Catanzaro, Calabria
  - Napoli, Campania
  - Rome, Lazio
  - Milan, Lombardy
  - Vicenza, Veneto
- Oslo, Norway
- Karachi, Pakistan
- Poland (2):
  - Krakow
  - Warsaw
- Serbia (3):
  - Belgrade
  - Niš
  - Novi Sad
- South Africa (2):
  - Pretoria, Gauteng
  - Parktown
- Spain (6):
  - A Coruña, A Coruña
  - Barcelona, Barcelona
  - Santander, Cantabria
  - Jaén, Jaén
  - Oviedo, Principality of Asturias
  - Valencia, Valencia
- Sweden (3):
  - Gothenburg
  - Malmo
  - Karolinska Universitetssjukhuset i Solna, Stockholm
- Taiwan (3):
  - Taipei, Taipei
  - Changhua
  - Taipei
- Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Adana
  - Antalya
  - Izmir
- United Kingdom (4):
  - Dundee, Dundee City
  - Oxford, Oxfordshire
  - Sheffield, South Yorkshire
  - London

REFERENCES:
- [Result] Kitchen S, Katterle Y, Beckmann H, Maas Enriquez M. Chromogenic assay for BAY 81-8973 potency assignment has no impact on clinical outcome or monitoring in patient samples. J Thromb Haemost. 2016 Jun;14(6):1192-9. doi: 10.1111/jth.13322. Epub 2016 May 3. PMID 27002680
- [Result] Oldenburg J, Windyga J, Hampton K, Lalezari S, Tseneklidou-Stoeter D, Beckmann H, Maas Enriquez M. Safety and efficacy of BAY 81-8973 for surgery in previously treated patients with haemophilia A: results of the LEOPOLD clinical trial programme. Haemophilia. 2016 May;22(3):349-53. doi: 10.1111/hae.12839. Epub 2016 Mar 1. PMID 26931631
- [Derived] Saxena K, Lalezari S, Oldenburg J, Tseneklidou-Stoeter D, Beckmann H, Yoon M, Maas Enriquez M. Efficacy and safety of BAY 81-8973, a full-length recombinant factor VIII: results from the LEOPOLD I trial. Haemophilia. 2016 Sep;22(5):706-12. doi: 10.1111/hae.12952. Epub 2016 Jun 24. PMID 27339736
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from specialized hemophilia treatment centers.
Pre-assignment Details: 14 participants were enrolled in each of Arms 1 and 2 in Part A. Of these, 11 participants continued into each of Arms 3 and 4 in Part B. Arm 3 enrolled 20 and Arm 4 enrolled 21 additional participants who had not participated in Part A. Arm 5 enrolled 5 participants specifically for surgery in Part C who had not participated in Parts A or B.
Groups:
- Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ: Part B - Arm 3: Participants received IV injection of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay Potency Per European Pharmacopeia (CS/EP) for 6 months and then crossed over to study drug measured by Chromogenic Substrate Assay/Adjusted (CS/ADJ) to Label Potency for 6 months
- Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP: Part B - Arm 4:. Participants received IV injection of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay/Adjusted (CS/ADJ) to Label Potency for 6 months and then crossed over to study drug measured by Chromogenic Substrate Assay Per European Pharmacopeia (CS/EP) for 6 months
- Arm 5: Recombinant Factor VIII by CS/EP: Part C - Arm 5: Participants received a loading dose of approximately 50 IU/kg of BAY81-8973 before the first surgical incision followed by further treatment with BAY81-8973 according to surgical requirements for up to 3 weeks
- Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension: Participants received IV injections of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay Potency Per European Pharmacopeia (CS/EP) for 6 months and CS/ADJ for 6 months sequence according to randomization and up to 12 months (CS/EP) during extension
Period: Part A Treatment Period
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII by CS/EP | Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension
Started | 14 | 14 | 0 | 0 | 0 | 0
Participants Received Treatment | 14 | 14 | 0 | 0 | 0 | 0
Safety Population | 13 (One excluded because receiving Kogenate FS twice.) | 14 | 0 | 0 | 0 | 0
Completed | 14 | 14 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Follow up Period
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII by CS/EP | Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension
Started | 14 | 14 | 0 | 0 | 0 | 0
Completed | 14 | 14 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B Treatment Period
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII by CS/EP | Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension
Started | 0 | 0 | 31 (Enrolled 4 participants from Arm 1 and 7 participants from Arm 2) | 32 (Enrolled 7 participants from Arm 1 and 4 participants from Arm 2) | 0 | 0
Participants Received Treatment | 0 | 0 | 30 | 32 | 0 | 0
Completed | 0 | 0 | 29 | 32 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Period: Part B Follow up Period
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII by CS/EP | Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension
Started | 0 | 0 | 29 | 32 | 0 | 0
Completed | 0 | 0 | 29 | 32 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII by CS/EP | Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension
Started | 0 | 0 | 0 | 0 | 0 | 55
Completed | 0 | 0 | 0 | 0 | 0 | 43
Not Completed | 0 | 0 | 0 | 0 | 0 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — starting another study | 0 | 0 | 0 | 0 | 0 | 8
Not completed — non-compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Period: Part C Treatment Period
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII by CS/EP | Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension
Started | 0 | 0 | 0 | 0 | 5 | 0
Participants Received Treatment | 0 | 0 | 0 | 0 | 5 | 0
Completed | 0 | 0 | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C Follow up Period
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII by CS/EP | Arm 6: Recombinant Factor VIII (BAY81-8973) Part B + Extension
Started | 0 | 0 | 0 | 0 | 5 | 0
Completed | 0 | 0 | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 5: Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C: Participants received a loading dose of approximately 50 IU/kg of BAY81-8973 before the first surgical incision, followed by further treatment with BAY81-8973 according to surgical requirements for up to 3 weeks
- Total: Total of all reporting groups
Arm/Group | Arm 1: Recombinant Factor VIII (BAY81-8973) Then Kogenate FS | Arm 2: Kogenate FS Then Recombinant Factor VIII (BAY81-8973) | Arm 3: Recombinant Factor VIII by CS/EP Then by CS/ADJ | Arm 4: Recombinant Factor VIII by CS/ADJ Then by CS/EP | Arm 5: Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C | Total
Number analyzed (Participants) | 14 | 14 | 20 | 21 | 5 | 74
Age, Customized [Number; unit: Participants] — Part A based on pharmacokinetic (PK) analysis set; Parts B and C based on safety analysis set
  Participants
    Part A < 18 years | 1 | 4 | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part A =/> 18 years | 12 | 9 | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part B < 18 years | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 5 | 5 | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part B =/> 18 years | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 25 | 27 | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part C < 18 years | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part C =/> 18 years | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Number; unit: Participants] — Part A based on PK analysis set; Parts B and C based on safety analysis set
  Participants
    Part A - Female | 0 | 0 | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part A - Male | 13 | 13 | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part B - Female | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 0 | 0 | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part B - Male | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 30 | 32 | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part C - Female | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Part C - Male | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | NA — Data is not available because participants did not participate in this phase. | 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
Most recent treatment before enrolment in the study [Number; unit: Participants] — Parts A, B and C all based on safety analysis set
  Participants
    On-demand | 4 | 3 | 4 | 8 | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Prophylaxis | 10 | 11 | 26 | 24 | NA — Data is not available because participants did not participate in this phase. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Part A - Area Under the Drug Concentration-time Curve (AUC)
Description: To examine the Pharmacokinetic (PK) characteristics of BAY 81-8973 and ensure that the new drug is similar to Kogenate FS. All results are based on the chromogenic assay.
Time Frame: Samples taken at pre-injection, and at 0.25, 0.5, 1, 3, 6, 8, 24, 30 and 48 hours post injection. AUC calculated from time of injection to infinity.
Population: PK Analysis Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Int.units x hours/deciliters (IU*h/dL)
Groups:
- Recombinant Factor VIII (BAY81-8973) - Part A: Participants received one single intravenous (IV) injection of BAY81-8973 50 IU/kg
- Kogenate FS (BAY14-2222) - Part A: Participants received one single intravenous (IV) injection of Kogenate FS (BAY14-2222) 50 IU/kg
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part A | Kogenate FS (BAY14-2222) - Part A
Number analyzed (Participants) | 26 | 26
Int.units x hours/deciliters (IU*h/dL) | 1889.23 (36.11) | 1583.91 (39.89)

2. Primary Outcome: Part A - Half-life (t 1/2)
Description: To examine the PK characteristics of BAY81-8973 and ensure that the new drug is similar to Kogenate FS. All results are based on the chromogenic assay.
Time Frame: Samples taken at pre-injection, and at 0.25, 0.5, 1, 3, 6, 8, 24, 30 and 48 hours post injection.
Population: PK Analysis Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part A | Kogenate FS (BAY14-2222) - Part A
Number analyzed (Participants) | 26 | 26
Hours (h) | 13.77 (28.00) | 12.00 (28.20)

3. Primary Outcome: Part B - Annualized Number of Total Bleeds
Description: The annualized number of bleeds experienced by participants
Time Frame: 12 months after randomization
Population: Intent to treat (ITT)
Measure: Median (Inter-Quartile Range); unit: Bleeds
Groups:
- Recombinant Factor VIII (BAY81-8973) - Part B: Participants received IV injections of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay Potency Per European Pharmacopeia (CS/EP) for 6 months and by Chromogenic Substrate Assay/Adjusted to Label Potency (CS/ADJ) for 6 months, sequence according to randomization.
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part B
Number analyzed (Participants) | 62
Bleeds | 1.03 [0.0 to 5.09]

4. Secondary Outcome: Part B - The in Vivo Recovery Values of Human Factor VIII (FVIII)
Description: The amount of Factor VIII found in blood samples taken after the injection of the study drug at the beginning of the CS/EP treatment period.
Time Frame: 15-30 minutes after the injection
Population: ITT. 1 measurement was taken in all participants at the start of the CS/EP labelled treatment period (CS/ADJ labelled treatment was experimental and will not be used for the future commercial drug, so no measurements were taken). Note: Only 59 of the 62 participants had valid recovery data.
Measure: Median (Inter-Quartile Range); unit: Kg/dL
Groups:
- Recombinant Factor VIII (BAY81-8973) by CS/EP - Part B: Participants received IV injections of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay Potency Per European Pharmacopeia (CS/EP) for 6 months
Arm/Group | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part B
Number analyzed (Participants) | 59
Kg/dL | 2.50 [2.09 to 2.77]

5. Secondary Outcome: Part B - Annualized Number of Bleeds in Each 6-month Potency Assignment Period
Description: The annualized number of bleeds experienced by participants in each of the two treatment periods
Time Frame: 6 months on each potency
Population: ITT. Note: One participant in Part B did not receive any Recombinant Factor VIII measured by the CS/ADJ method, leading to 61 participants (not 62) in that group.
Measure: Median (Inter-Quartile Range); unit: Bleeds
Groups:
- Recombinant Factor VIII (BAY81-8973) by CS/ADJ - Part B: Participants received IV injection of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay/Adjusted (CS/ADJ) to Label Potency for 6 months
Arm/Group | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part B | Recombinant Factor VIII (BAY81-8973) by CS/ADJ - Part B
Number analyzed (Participants) | 62 | 61
Bleeds | 1.9 [0.0 to 4.4] | 1.9 [0.0 to 7.3]

6. Secondary Outcome: Part B - Control of Bleeding as Measured by the Number of Injections Required to Treat a Bleed
Description: The number of injections needed by participants to stop a bleed
Time Frame: 6 months on each potency
Population: as for outcome 5
Measure: Median (Full Range); unit: Injections
Units Other Than Participants: Bleeds
Arm/Group | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part B | Recombinant Factor VIII (BAY81-8973) by CS/ADJ - Part B
Number analyzed (Participants) | 62 | 61
Number analyzed (Bleeds) | 108 | 128
Injections | 1.0 [0 to 11] | 1.0 [1 to 48]

7. Secondary Outcome: Part B - Changes From Baseline at 12 Months in Quality of Life (QoL) as Measured by Transformed Total Score of Haemo-QoL Questionnaire
Description: A measure of how treatment with BAY81-8973 affected the daily life of participants. the scoring system has 100 points. 0 is the worst possible score. 100 is the best possible score. Positive changes from baseline indicate an improvement in quality of life and negative changes indicate a deterioration.
Time Frame: Baseline and 12 months
Population: ITT. Note: Only 51 of the 62 participants had data available for the 12-month QoL analysis.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part B
Number analyzed (Participants) | 51
Scores on a scale | 2.02 [-22.9 to 26.5]

8. Secondary Outcome: Part B - Changes From Baseline at 12 Months in Utility Index as Measured by EQ-5D Questionaire
Description: A measure of how treatment with BAY81-8973 affected the daily life of participants. 1.0 = Best possible score, -0.594 = Worst possible score. Positive changes from baseline indicate an improvement and negative changes indicate a deterioration.
Time Frame: Baseline and 12 months
Population: ITT. Note: Only 61 of the 62 participants had data available for the Utility Index of the EQ-5D questionnaire at Month 12.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part B
Number analyzed (Participants) | 61
Scores on a scale | 0.00 [-0.6 to 0.5]

9. Secondary Outcome: Part A - Number of Participants With Inhibitory Antibody Formation
Description: A test to ensure that participants have not developed antibodies that will interfere with the action of BAY81-8973
Time Frame: Up to 6 weeks after first injection of study drug
Population: Safety population
Measure: Number; unit: Participants
Groups:
- Recombinant Factor VIII (BAY81-8973) and Kogenate FS - Part A: Participants received one single intravenous (IV) injection of BAY81-8973 50 IU/kg and one single intravenous (IV) injection of Kogenate FS (BAY14-2222) 50 IU/kg
Arm/Group | Recombinant Factor VIII (BAY81-8973) and Kogenate FS - Part A
Number analyzed (Participants) | 28
Participants | 0

10. Secondary Outcome: Part B - Number of Participants With Incidence of Inhibitory Antibody Formation
Description: A test to ensure that participants have not developed antibodies that will interfere with the action of BAY81-8973
Time Frame: Up to 12 months after drug administration
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part B
Number analyzed (Participants) | 62
Participants | 0

11. Secondary Outcome: Part C - Number of Participants With Incidence of Inhibitory Antibody Formation
Description: A test to ensure that participants have not developed antibodies that will interfere with the action of BAY81-8973
Time Frame: before and 3 weeks after surgery
Population: ITT
Measure: Number; unit: Participants
Groups:
- Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C: Participants received a loading dose of approximately 50 IU/kg of BAY81-8973 before the first surgical incision, followed by further treatment with BAY81-8973 according to surgical requirements for up to 3 weeks
Arm/Group | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C
Number analyzed (Participants) | 5
Participants | 0

12. Secondary Outcome: Part A - Number of Participants With Incidence of Antibody Formation to Heat-shock Protein (HSP-70)
Description: A test to analyze the formation of antibodies to HSP-70
Time Frame: Up to 6 weeks after drug administration
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) and Kogenate FS - Part A
Number analyzed (Participants) | 28
Participants | 0

13. Secondary Outcome: Part B - Number of Participants With Incidence of Antibody Formation to Heat-shock Protein (HSP-70)
Description: A test to analyze the formation of antibodies to HSP-70
Time Frame: Up to 12 months after drug administration
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part B
Number analyzed (Participants) | 62
Participants | 1

14. Secondary Outcome: Part C - Number of Participants With Incidence of Antibody Formation to Heat-shock Protein (HSP-70)
Description: A test to analyze the formation of antibodies to HSP-70
Time Frame: before and 3 weeks after surgery
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C
Number analyzed (Participants) | 5
Participants | 0

15. Secondary Outcome: Part A - Number of Participants With Incidence of Antibody Formation to Host Cell Proteins (HCP)
Description: A test to ensure that participants have not developed antibodies to HCP during the study
Time Frame: Up to 4 weeks after drug administration
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) and Kogenate FS - Part A
Number analyzed (Participants) | 26
Participants | 0

16. Secondary Outcome: Part B - Number of Participants With Incidence of Antibody Formation to Host Cell Proteins (HCP)
Description: A test to ensure that participants have not developed antibodies to HCP during the study
Time Frame: Up to 12 months after drug administration
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part B
Number analyzed (Participants) | 62
Participants | 0

17. Secondary Outcome: Part C - Number of Participants With Incidence of Antibody Formation to Host Cell Proteins (HCP)
Description: A test to ensure that participants have not developed antibodies to HCP during the study
Time Frame: before and 3 weeks after surgery
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C
Number analyzed (Participants) | 5
Participants | 0

18. Secondary Outcome: Part B - Number of Participants With Assessment of the Hemostasis During Major Surgery
Description: An assessment made by surgeons of how effective BAY81-8973 was in stopping bleeding during major operations
Time Frame: An average of 1 month after start of treatment
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part B
Number analyzed (Participants) | 5
Participants
  Excellent | 1
  Good | 4
  Moderate | 0
  Poor | 0

19. Secondary Outcome: Part C - Number of Participants With Assessment of the Hemostasis During Major Surgery
Description: An assessment made by surgeons of how effective BAY81-8973 was in stopping bleeding during major operations
Time Frame: at the time of surgery
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C
Number analyzed (Participants) | 5
Participants
  Excellent | 1
  Good | 4
  Moderate | 0
  Poor | 0

ADVERSE EVENTS:
Time Frame: From the date of signing informed consent through study completion, i.e. 21 Dec 2009 to 14 Mar 2013
Description: The objective of Part C was efficacy assessment of surgery hemostasis, not safety assessment. It was allowed to include the same patient for several surgeries and for each surgery the patient was assigned a new patient number. Due to this approach, one patient with 3 surgeries was analyzed as 3 different patients, therefore the number at risk is 7.
Groups:
- Recombinant Factor VIII (BAY81-8973) Part B and Extension: Participants received IV injections of BAY81-8973 at 20-50 IU/kg 2-3 times per week with BAY81-8973 measured by Chromogenic Substrate Assay Potency Per European Pharmacopeia (CS/EP) for 6 months and CS/ADJ for 6 months sequence according to randomization and up to 12 months (CS/EP) during extension
- Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C: Participants in Part C received a loading dose of approximately 50 IU/kg of BAY81-8973 (nearest whole vial amount) for less than 15 minutes before the first surgical incision. Then they received further treatment with BAY81-8973 according to surgical requirements up to 3 weeks.
Arm/Group | Recombinant Factor VIII (BAY81-8973) - Part A | Kogenate FS (BAY14-2222) - Part A | Recombinant Factor VIII (BAY81-8973) Part B and Extension | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 12/62 | 1/7
Other Adverse Events (participants affected / at risk) | 0/27 | 1/28 | 43/62 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Factor VIII (BAY81-8973) - Part A (N=27) | Kogenate FS (BAY14-2222) - Part A (N=28) | Recombinant Factor VIII (BAY81-8973) Part B and Extension (N=62) | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C (N=7)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2 | 0
Spinal pain (General disorders) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Somatoform disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Miscarriage of partner (Social circumstances) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Factor VIII (BAY81-8973) - Part A (N=27) | Kogenate FS (BAY14-2222) - Part A (N=28) | Recombinant Factor VIII (BAY81-8973) Part B and Extension (N=62) | Recombinant Factor VIII (BAY81-8973) by CS/EP - Part C (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thymus disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 4 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Chest pain (General disorders) | 0 | 0 | 4 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 0 | 6 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 14 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 8 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days